CLINICAL TRIAL: NCT03415126
Title: A Phase 1, Open-Label, Dose-Finding Study Of ASN007 In Patients With Advanced Solid Tumors
Brief Title: A Study of ASN007 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN007-101
Record Dates: First submitted 2018-01-15; First posted 2018-01-30 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Cancer; Malignancy; Neoplasia; Neoplasm; Neoplasm Metastasis; Colon Cancer; Colonic Neoplasms; Colon Cancer Liver Metastasis; Metastatic Cancer; Metastatic Melanoma; Metastatic Colon Cancer; Metastatic Lung Cancer; Non Small Cell Lung Cancer Metastatic; Pancreatic Cancer; Pancreas Cancer; Pancreas Adenocarcinoma; Pancreas Neoplasm; Metastatic Nonsmall Cell Lung Cancer; Metastatic Pancreatic Cancer
Keywords: KRAS mutant; NRAS mutant; BRAF mutant; HRAS mutant; ERK 1/2 inhibitor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Melanoma; Lung Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- ASN007 ascending doses (Experimental): Patients will receive escalating doses of ASN007 to identify the best dose.
  Interventions: Drug: ASN007: ascending doses
- ASN007 RD: KRAS mutant Melanoma (Experimental): Patients with BRAF mutant metastatic melanoma will receive the recommended dose from Part A.
  Interventions: Drug: ASN007 RD
- ASN007 RD: NRAS mutant Melanoma (Experimental): Patients with NRAS and HRAS mutant solid tumors will receive the recommended dose from Part A.
  Interventions: Drug: ASN007 RD
- ASN007 RD: KRAS mutant metastatic CRC (Experimental): Patients with KRAS mutant CRC will receive the recommended dose from Part A
  Interventions: Drug: ASN007 RD
- ASN007 RD: KRAS mutant NSCLC (Experimental): Patients with KRAS mutant NSCLC will receive the recommended dose from Part A
  Interventions: Drug: ASN007 RD
- ASN007 RD: Metastatic Pancreatic Cancer (Experimental): Patients with pancreatic adenocarcinoma will receive the recommended dose from Part A
  Interventions: Drug: ASN007 RD
- ASN007 RD: MEK, All BRAF, BRAF-fusion cancers (Experimental): Patients with solid tumors will receive the recommended dose from Part A
  Interventions: Drug: ASN007 RD

INTERVENTIONS:
Drug: ASN007: ascending doses — Oral drug for the treatment of advanced solid tumors
  Arms: ASN007 ascending doses
Drug: ASN007 RD — Oral drug for the treatment of advanced solid tumors
  Arms: ASN007 RD: KRAS mutant Melanoma; ASN007 RD: KRAS mutant NSCLC; ASN007 RD: KRAS mutant metastatic CRC; ASN007 RD: MEK, All BRAF, BRAF-fusion cancers; ASN007 RD: Metastatic Pancreatic Cancer; ASN007 RD: NRAS mutant Melanoma

SUMMARY:
The study is divided into two parts. The first part of the study will test various doses of ASN007 to find out the highest safe dose to test in five specific groups. The second part of the study will test how well ASN007 can control cancer.

DETAILED DESCRIPTION:
Part A is a dose escalation study to determine a safe and tolerable dose of ASN007 for patients with advanced solid tumors. Part A will also describe how the body works on ASN007(pharmacokinetics) and the effects of ASN007 on the body (pharmacodynamics) of ASN007, through blood sampling and optional biopsies..

Part B of the study will enroll patients with particular tumor types and genetic mutations for treatment at the Recommended Phase 2 Dose. Part B will enroll patients in five groups of fifteen patients each:

Group 1: Patients with metastatic BRAF mutated melanoma Group 2: Patients with metastatic NRAS and HRAS mutated solid tumors Group 3: Patients with metastatic KRAS mutated colorectal cancer (CRC) Group 4: Patients with metastatic KRAS mutated non-small cell lung cancer (NSCLC) Group 5: Patients with metastatic pancreatic ductal adenocarcinoma (PDAC) Patients with melanoma will be required to have pre-dose and post-dose biopsies.

Group 6: Patients with metastatic MEK1, BRAF V600E, non-BRAF V600E solid tumors or BRAF fusions without prior treatment with BRAF, MEK, ERK inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-related procedure being performed;
* Male or non-pregnant, non-lactating female patient at least 18 years of age at the time of consent;
* Eastern Cooperative Oncology Group Performance Status 0-1 (Part A) and PS 0-2 (Part B)
* Histologically or cytologically confirmed
* advanced or metastatic solid tumor (Part A)
* Group 1: BRAF mutant melanoma (Part B)
* Group 2: NRAS or HRAS mutant solid tumors(Part B)
* Group 3: KRAS mutant CRC.(Part B)
* Group 4: KRAS mutant NSCLC (Part B)
* Group 5: Pancreatic Ductal Adenocarcinoma (Part B)
* Progressive disease after failure of or intolerant to all available standard systemic treatments that have shown a documented benefit in overall survival for their respective tumor type.
* Measurable or evaluable disease per RECIST v1.1
* Screening hematology values of the following:
* absolute neutrophil count ≥ 1000/μL,
* platelets ≥ 100,000/μL,
* hemoglobin ≥ 9 g/dL
* Screening chemistry values of the following:
* alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3.0 × upper limit of the normal (ULN),
* total bilirubin ≤ 1.5 × ULN,
* creatinine ≤ 1.5 × ULN,,
* albumin ≥ 2.8 g/dL.
* Screening heart function lab test
* creatinine kinase - MB, troponin-I, and troponin-T within normal limits
* Subject is willing and able to comply with all protocol required visits and assessments, including biopsy if assigned.

Exclusion Criteria:

* Prior treatment with ASN007 or another ERK1/2 inhibitor
* Known hypersensitivity to ASN007 or its excipients;
* Part B: Prior treatment with a RAF or MEK pathway inhibitor, except BRAFmutant melanoma (Group 1)
* Prior chemotherapy, targeted therapy or monoclonal antibody therapy within 3 weeks of start of study treatment (Day1), or 5 half-lives, whichever is shorter.
* Concurrent or prior bone marrow factors (e.g. G-CSF, GM-CSF or erythropoietin) within 3 weeks prior to Day 1 of treatment.
* Febrile neutropenia or serious persistent infection within 2 weeks prior to Day 1 of treatment
* Failure to recover from major surgery or traumatic injury within 4 weeks or minor surgery within 2 weeks prior to Day 1 of treatment.
* History of or current evidence / risk of retinal vein occlusion (RVO) central serous retinopathy (CSR), or glaucoma with intraocular pressures ≥ 21 mmHg or other pre-existing ocular conditions that may put the patient at risk for ocular toxicities
* Known central nervous system (CNS) primary tumor, CNS metastases or carcinomatous meningitis (Part A). Patients may be enrolled with CNS metastasis in certain circumstances in Part B.
* Clinically significant heart disorders including an ejection fraction of < 50%
* Other serious uncontrolled conditions such as fungal, bacterial or viral infection; HIV, Hepatitis B or C, bleeding disorders, interstitial lung disease,
* Any other condition that might place the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Part A: Determine the maximum tolerated dose (MTD) of ASN007 | First 21 days
  The MTD will be determined by evaluating the number of subjects with treatment related dose limiting toxicity. This is the primary endpoint of Part A
Part B: evaluate the overall response rate (number of Complete Responses + Partial Responses) in subjects receiving ASN007 for the treatment of metastatic melanoma, CRC, NSCLC, or pancreatic cancer. | First 6 months
  This is the primary endpoint for Part B.

SECONDARY OUTCOMES:
Calculate the pharmacokinetic area under the plasma concentration (AUC) of ASN007 | First 21 days
  Calculate the amount of ASN007 in the bloodstream
Calculate the maximum plasma concentration (Cmax) at steady state. | First 21 days
  Calculate the maximum amount of ASN007 in the bloodstream
Calculate the terminal elimination rate (T 1/2). | First 21 days
  Calculate how fast ASN007 leaves the body

OTHER OUTCOMES:
To evaluate the change from baseline in the intensity of phosphorylated ribosomal S6 kinase (RSK) found in tumor biopsies. | Through the study, average 6 months
  Evaluate the effect of ASN007 on biomarkers
Evaluate the change from baseline in the amount of circulating tumor DNA | Every 8 weeks for the first 24 weeks, then every 12 weeks for up to 1 year
  Evaluate the effect of ASN007 on biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Asana BioSciences
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No